CLINICAL TRIAL: NCT03020251
Title: Effects of Preoperative Rehabilitation in Patients Resected for Lung Cancer
Acronym: Rexochir
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-A00622-49
Record Dates: First submitted 2016-12-20; First posted 2017-01-13 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Lungcancer
Keywords: preoperative rehabilitation program; chest physiotherapy; lung cancer resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (C group) (Active Comparator): patient will receive preoperative chest physiotherapy (standard supportive care)
  Interventions: Other: preoperative chest physiotherapy
- rehabilitation group (R group) (Experimental): patient will receive preoperative chest physiotherapy and a preoperative rehabilitation program at home (exercise training)
  Interventions: Other: preoperative chest physiotherapy; Other: preoperative rehabilitation program

INTERVENTIONS:
Other: preoperative chest physiotherapy — preoperative chest physiotherapy : 5 sessions per week during 3 weeks
Other: preoperative rehabilitation program — exercise training at home : 5 sessions per week during 3 weeks
  Arms: rehabilitation group (R group)

SUMMARY:
This randomized controlled trial will evaluate the effect of a preoperative rehabilitation program at home in patients resected for lung cancer, comparing a control group (C group) receiving only chest physiotherapy and a rehabilitation group (R group) receiving both a training program at home and chest physiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed for lung cancer (or highly suspicious for cancer tumor) eligible for resection surgery (lobectomy or pneumonectomy)
* Age > 18 years
* Presence of Chronic Obstructive Pulmonary Disease (COPD) stages 2-4 of Gold (forced expiratory volume (FEV )/ forced vital capacity (FVC) <70%, FEV <80% of predicted) and Exertional dyspnea stage MMRC (Medical Research Council) > 1
* Patients must provide written consent
* Member of social security scheme

Exclusion Criteria:

* Patients refusing to participate
* COPD stage 1 Gold (VEMS >= 80% of the theoretical value)
* Presenting an operating contraindication during the initial maximal exercise test
* Presenting cardiac or vascular contraindication to achieve the readaptation program
* Patient living alone at home
* Patient with ventilatory assistance at home (oxygen therapy or noninvasive ventilation (NIV))
* With exercise hypoventilation (PaCO2 >45 mmHg)
* Cognitive difficulty
* unable major
* pregnancy,
* patients deprived of liberty by a court or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-05-12 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay after resection for lung cancer | time from the date of the surgery (Day 0) until the date of discharge (Day n) (assessed up to 56 days)
  the date of discharge will be the real day of discharge from surgery department or the day where the patient will be medically considered as outgoing

SECONDARY OUTCOMES:
the number of complications | during the stay in the surgery department or the intensive care unit (up to 56 days)
peak oxygen consumption | evaluation N°1 : during the week before the first date of the intervention (week 1). evaluation N°2: during the week before the date of surgery (week 5)
  evaluation N°1 before intervention : during the week before the first date of the intervention (week 1) (intervention : preoperative chest physiotherapy +/- rehabilitation program will be realized on weeks 2, 3, and 4).
  evaluation N°2 after intervention and before surgery : during the week before the date of surgery (week 5)
6 minutes walking distance | evaluation N°1 : during the week before the first date of the intervention (week 1). evaluation N°2: during the week before the date of surgery (week 5)
  evaluation N°1 before intervention : during the week before the first date of the intervention (week 1) (intervention : preoperative chest physiotherapy +/- rehabilitation program will be realized on weeks 2, 3, and 4).
  evaluation N°2 after intervention and before surgery : during the week before the date of surgery (week 5)
maximal voluntary quadriceps strength | evaluation N°1 : during the week before the first date of the intervention (week 1). evaluation N°2: during the week before the date of surgery (week 5)
  evaluation N°1 before intervention : during the week before the first date of the intervention (week 1) (intervention : preoperative chest physiotherapy +/- rehabilitation program will be realized on weeks 2, 3, and 4).
  evaluation N°2 after intervention and before surgery : during the week before the date of surgery (week 5)
maximal inspiratory and expiratory strength | evaluation N°1 : during the week before the first date of the intervention (week 1). evaluation N°2: during the week before the date of surgery (week 5)
  evaluation N°1 before intervention : during the week before the first date of the intervention (week 1) (intervention : preoperative chest physiotherapy +/- rehabilitation program will be realized on weeks 2, 3, and 4).
  evaluation N°2 after intervention and before surgery : during the week before the date of surgery (week 5)
real length of stay | between the first postoperative day (Day 1) and the real discharge date (up to 56 days)
  the real day of discharge from surgery department
body composition (bioimpedancemetry) | evaluation N°1 : during the week before the first date of the intervention (week 1). evaluation N°2: during the week before the date of surgery (week 5)
  evaluation N°1 before intervention : during the week before the first date of the intervention (week 1) (intervention : preoperative chest physiotherapy +/- rehabilitation program will be realized on weeks 2, 3, and 4).
  evaluation N°2 after intervention and before surgery : during the week before the date of surgery (week 5)
oxidative adaptations of the muscle | evaluation N°1 : during the week before the first date of the intervention (week 1). evaluation N°2 after intervention : at the date of surgery (during the surgical time at Day 0 week 6)
  optional ancillary study on quadricipal and intercostal muscle biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Marc FILAIRE, Pr, Principal Investigator — Centre Jean Perrin
Locations (6):
- France (6):
  - CHU Clermont Ferrand, Gabriel Montpied, service de médecine du sport et explorations fonctionnelles,, Clermont-Ferrand
  - Centre de Recherche en Nutrition Humaine, Clermont-Ferrand
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU Grenoble, Hôpital Michallon, Grenoble
  - Hospices Civiles de Lyon, groupement hospitalier Est, Hopital Louis Pradel, Lyon
  - CHU Saint-Etienne, CHU Hopital Nord, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laurent H, Galvaing G, Thivat E, Coudeyre E, Aubreton S, Richard R, Kwiatkowski F, Costes F, Filaire M. Effect of an intensive 3-week preoperative home rehabilitation programme in patients with chronic obstructive pulmonary disease eligible for lung cancer surgery: a multicentre randomised controlled trial. BMJ Open. 2017 Nov 12;7(11):e017307. doi: 10.1136/bmjopen-2017-017307. PMID 29133320